CLINICAL TRIAL: NCT02391870
Title: Phase One: An Open Trial of Mindfulness-Based Cognitive Therapy for the Prevention of Perinatal Depression
Brief Title: The Staying Well Study: An Open Trial of Mindfulness-Based Cognitive Therapy for the Prevention of Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Emory University (Other); Kaiser Permanente (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sona Dimidjian, Professor and Director, University of Colorado, Boulder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-0353-01; R34MH083866 (NIH)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Pregnancy; Depression; Postpartum Depression
Keywords: depression; mindfulness; pregnancy; prevention; cognitive behavioral therapy
MeSH Terms: conditions — Depression; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MBCT-PD (Experimental): Mindfulness-based cognitive therapy adapted for perinatal women (MBCT-PD)
  Interventions: Behavioral: MBCT-PD

INTERVENTIONS:
Behavioral: MBCT-PD — Using an iterative process, the investigators modified MBCT to include a focus on perinatal depression (MBCT-PD). The modifications took into account developmental processes associated with the perinatal period, characteristics and correlates of perinatal depression, and the physical aspects of pregnancy.

SUMMARY:
Pregnant women with histories of depression are at high risk of depressive relapse during the perinatal period, and options for relapse prevention are limited. Mindfulness-based cognitive therapy (MBCT) has strong evidence among general populations but has not been studied among at risk pregnant women.

This study is the first phase of a multi-phase project adapting MBCT for perinatal women (MBCT-PD). It is being conducted in a collaboration between the University of Colorado, Emory University, and Kaiser Permanente at Colorado and Georgia.

DETAILED DESCRIPTION:
Mindfulness-based cognitive therapy (MBCT) represents one of the most important recent developments in the effort to prevent recurrent depression. Explicitly designed to modify core underlying vulnerability factors among recovered individuals with histories of depression, MBCT may have high applicability to the prevention of perinatal depression (PD).

During this phase of the project the investigators will employ an iterative process to develop, within routine obstetric clinical settings, the MBCT-PD program across a two-center open trial of pregnant women at high risk of perinatal depression. During this phase, the investigators will modify the standard MBCT approach to be sensitive and specific to women at high risk of perinatal depressive relapse or recurrence based on previous history of depression and will address the following aims:

* Specific Aim 1: To examine the feasibility of MBCT-PD with respect to identification and enrollment of women at-risk of perinatal depression based on a history of depression.
* Specific Aim 2: To examine the engagement of women with the MBCT-PD approach with respect to retention, completion of daily practice assignments, and satisfaction
* Specific Aim 3: To examine the clinical outcomes including change in depression symptom levels and rates of relapse/recurrence over the course of the intervention and through a 6-month postpartum follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant up to 32 weeks gestation
* Meeting criteria for prior depression
* Failure to meet criteria for a diagnosis of MDD in the last two months
* Available for group intervention scheduled meetings

Exclusion Criteria:

* Presence of schizophrenia or schizoaffective disorder
* Presence of bipolar disorder or current psychosis
* Presence of organic mental disorder or pervasive developmental delay
* Presence of current eating disorder
* Presence of current substance abuse or dependence
* Presence of antisocial, borderline, or schizotypal personality disorder
* Presence of imminent suicide or homicide risk
* Presence of any other axis I or II disorders that necessitate priority treatment not provided by the study protocol
* Women with any medical conditions that would preclude participation, including high-risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Engagement | Up to 8 weeks
  Engagement is operationalized in-part as class attendance, with completion is defined as attendance at a minimum of four classes, and daily home practice recorded daily as the number of times of practice and type of practice, which are classified as either formal or informal practice.
Client Satisfaction | Up to 8 weeks
  Participant satisfaction will be evaluated by the CSQ-8, which is designed to yield a homogeneous estimate of general satisfaction with services. An exit interview also will be completed at 6-months postpartum.
MBCT-PD Adherence Scale (MBCT-PD-AS) | Up to 8 weeks
  Treatment fidelity will be assessed to provide checks on the adequacy of treatment implementation, using the MBCT-PD Adherence Scale.
Depressive Relapse Status: Longitudinal Interval Follow-up Evaluation (LIFE) | Up to 6 months postpartum
  Rate of depressive relapse and time to relapse will be assessed using the LIFE, which provides a retrospective assessment of relapse or recurrence based on a semi-structured interview according to DSM-IV-TR diagnostic criteria.
Change in Edinburgh Postpartum Depression Scale (EPDS) | Up to 6 months postpartum
  Change in the severity of depressive symptoms will be evaluated by the Edinburgh Postpartum Depression Scale (EPDS), which is the most widely used self-report measure of antenatal and postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sona Dimidjian, PhD, Principal Investigator — University of Colorado, Boulder; Sherryl Goodman, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - University of Colorado Boulder, Boulder, Colorado
  - Kaiser Permanente Colorado, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Kaiser Permanente, Atlanta, Georgia